CLINICAL TRIAL: NCT00129766
Title: A Pivotal Phase 3 Study of MEDI-524 (Numax; Motavizumab), an Enhanced Potency Humanized RSV Monoclonal Antibody, for the Prophylaxis of Serious RSV Disease in High-Risk Children
Brief Title: Study of MEDI-524 (Motavizumab) for the Prophylaxis of Serious Respiratory Syncytial Virus (RSV) Disease in High-Risk Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MI-CP110
Record Dates: First submitted 2005-08-10; First posted 2005-08-12 (Estimated); Results first posted 2013-08-28 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-06

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Respiratory Syncytial Virus (RSV); motavizumab; palivizumab; Synagis
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — motavizumab; Palivizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- palivizumab (Active Comparator): 15 mg/kg administered intramuscularly for 5 monthly doses
  Interventions: Biological: palivizumab
- motavizumab (MEDI-524) (Experimental): 15 mg/kg of motavizumab was administered intramuscularly for 5 monthly doses
  Interventions: Biological: motavizumab (MEDI-524)

INTERVENTIONS:
Biological: motavizumab (MEDI-524) — Motavizumab, 15 mg/kg administered intramuscularly for 5 monthly doses
  Other Names: MEDI-524
  Arms: motavizumab (MEDI-524)
Biological: palivizumab — Palivizumab, 15 mg/kg administered intramuscularly for 5 monthly doses
  Other Names: Synagis
  Arms: palivizumab

SUMMARY:
The primary objective of this study was to compare the safety and efficacy of motavizumab to palivizumab when administered monthly by intramuscular (IM) injection for the reduction of the incidence of RSV hospitalization among children at high risk for serious RSV disease. A secondary objective was to compare the incidence of medically-attended lower respiratory infections (LRIs) between treatment groups.

DETAILED DESCRIPTION:
A randomized, double-blind, palivizumab-controlled, multi-center, multi-national trial conducted during 2 Northern Hemisphere RSV seasons with an intervening season in the Southern Hemisphere. Each child only participated during a single RSV season. Approximately 6,600 children at risk for serious RSV disease were to be randomized in a 1:1 ratio to receive either 15 mg/kg of palivizumab or motavizumab by IM injection every 30 days for a total of 5 doses.

ELIGIBILITY:
Inclusion Criteria:

* 24 months of age or younger at randomization (child must be randomized on or before his/her 24-month birthday) with a diagnosis of chronic lung disease (CLD) of prematurity requiring medical intervention/management (i.e., supplemental oxygen, bronchodilators, or diuretics) within 6 months before randomization

OR:

* 35 weeks gestational age or less at birth and 6 months of age or younger at randomization (children were to be randomized on or before his/her 6-month birthday)

Exclusion Criteria:

* Hospitalization at the time of randomization (unless discharge was anticipated within 10 days)
* Mechanical ventilation or other mechanical support (including continuous positive airways pressure [CPAP])
* Life expectancy < 6 months
* Active RSV infection (a child with signs/symptoms of respiratory infection must have had negative RSV testing)
* Known renal impairment
* Known hepatic dysfunction
* Chronic seizure or evolving or unstable neurologic disorder
* Congenital heart disease [CHD] (children with uncomplicated CHD [e.g., patent ductus arterious (PDA), small septal defect] and children with complicated CHD that were currently anatomically and hemodynamically normal could be enrolled)
* Known immunodeficiency
* Mother with HIV infection (unless the child has been proven to be not infected)
* Known allergy to Ig products
* Receipt of palivizumab, RSV-IGIV, or other RSV-specific monoclonal antibody, or any other polyclonal antibody (for example, hepatitis B IG, IVIG, VZIG) within 3 months prior to randomization
* Anticipated use of palivizumab or IVIG during the study (blood transfusions permitted)
* Previous receipt of RSV vaccines
* Participation in other investigational drug product studies

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6635 (Actual)
Dates: Start 2004-11; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M Pamela Griffin, MD, Study Director — MedImmune LLC
Locations (343):
- United States (120):
  - University Of Alabama At Birmingham, Birmingham, Alabama
  - Alabama Neonatal Medicine OC, Pike Road, Alabama
  - Maricopa Medical Center, Phoenix, Arizona
  - Central Arkansas Pediatric Clinic, PA, Benton, Arkansas
  - The Children's Clinic Of Jonesboro, P.A., Jonesboro, Arkansas
  - Arkansas Children's Hospital Research Institute, Little Rock, Arkansas
  - Arkansas Pediatric Clinic, Little Rock, Arkansas
  - Little Rock Children's Clinic, PA, Little Rock, Arkansas
  - Miller Children's Hospital, Long Beach, California
  - Kaiser Permanente Los Angeles, Los Angeles, California
  - Children's Hospital of Oakland, Oakland, California
  - Kaiser Permanente Health Care Plan, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - University of California, San Diego, California
  - Children's Hospital San Diego, San Diego, California
  - California Pacific Medical Center, San Francisco, California
  - Santa Clara Valley Medical Center, San Jose, California
  - Children's Hospital, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Pediatric Pulmonology, LLC, Stamford, Connecticut
  - A. I. Dupont Hospital For Children, Wilmington, Delaware
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Shands Hospital At The University Of Florida, Gainesville, Florida
  - The Nemours Children's Clinic, Jacksonville, Florida
  - University Of Miami Medical Center, Miami, Florida
  - Nemours Children's Clinic Biomedical Research, Orlando, Florida
  - Univ. S. Florida Pediatrics Ambulatory Care Center, Tampa, Florida
  - Emory University School Of Medicine, Atlanta, Georgia
  - Georgia Pediatric Pulmonology Associates, Atlanta, Georgia
  - The Medical College Of Georgia, Augusta, Georgia
  - Kapiolani Medical Center for Woman and Children, Honolulu, Hawaii
  - University of Illinois at Chicago, Chicago, Illinois
  - Children's Memorial Hospital, Chicago, Illinois
  - Advocate Hope Children's Hospital, Cook, Illinois
  - Lutheran General Children's Hospital, Park Ridge, Illinois
  - James Whitcomb Riley Hospital for Children, Indianapolis, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - University of Louisville, Louisville, Kentucky
  - Louisiana State University MidCity Clinic, Baton Rouge, Louisiana
  - Tulane Hospital for Children, New Orleans, Louisiana
  - University Of Maryland School of Medicine, Baltimore, Maryland
  - Tufts-New England Medical Center, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Michigan Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital Of Michigan, Detroit, Michigan
  - St. John Hospital & Medical Center, Detroit, Michigan
  - DeVos Children's Hospital, Grand Rapids, Michigan
  - St. Mary's Duluth Clinic, Duluth, Minnesota
  - Children's Healthcare D.B.A. Hospitals & Clinics, Saint Paul, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - University of Nebraska Medical Center Pediatric, Omaha, Nebraska
  - Children's Lung Specialist, Ltd, Las Vegas, Nevada
  - Dartmouth Medical School, Lebanon, New Hampshire
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - New Jersey Medical School, Newark, New Jersey
  - Albany Medical Center, Albany, New York
  - The Brooklyn Hospital Center, Brooklyn, New York
  - Women & Children's Hospital, Buffalo, New York
  - Winthrop University Hospital, Mineola, New York
  - Schneider Children's Hospital, New Hyde Park, New York
  - The Children's Medical Group, Poughkeepsie, New York
  - University Of Rochester Medical Center, Rochester, New York
  - University Hospital State University of New York at Stony Brook Department of Pediatrics, Stony Brook, New York
  - Crouse Hospital NICU, Syracuse, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Bronx-Lebanon Hospital Center, The Bronx, New York
  - Jacobi Medical Center, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina-School of Medicine, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University School of Medicine, Greenville, North Carolina
  - Raleigh Pediatric Associates, Raleigh, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Children's Hospital Medical Center Of Akron, Akron, Ohio
  - Beehly Medical Park Women's and Children's Pav., Boardman, Ohio
  - University of Cincinnati Col. of Med., Cincinnati, Ohio
  - Metro Health Medical Center, Cleveland, Ohio
  - Pediatric Clinical Trials International, Inc., Columbus, Ohio
  - Children's Medical Center, Dayton, Ohio
  - Tod Children's Hospital, Mahaning, Ohio
  - Toledo Children's Hospital, Toledo, Ohio
  - St. Vincent Medical Center, Toledo, Ohio
  - Children's Hospital Of Oklahoma, Oklahoma City, Oklahoma
  - Saint Francis Hospital EOPC, Tulsa, Oklahoma
  - Oregon Health Sciences University, Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - St. Luke's Hospital, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center- JW Children's Hospital, Danville, Pennsylvania
  - The Children's Hospital Of Philadelphia, Philadelphia, Pennsylvania
  - Jefferson-duPont Children's Health Program, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - MUSC, Charleston, South Carolina
  - Sioux Valley Hospital University of South Dakota Medical Center, Sioux Falls, South Dakota
  - Lebonheur Children's Medical Center, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Baylor University Medical Center, Dallas, Texas
  - Univ. Of Texas Southwestern Medical Center, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - University Of Texas Houston Medical School, Houston, Texas
  - Texas Tech Health Sciences Center, Lubbock, Texas
  - University Of Texas Health Science Center, San Antonio, Texas
  - Scott & White Memorial Hospital, Temple, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - University of Virginia Hospital, Charlottesville, Virginia
  - VCU Medical Center, Richmond, Virginia
  - University Physicians, Huntington, West Virginia
  - West Virginia University, Morgantown, West Virginia
  - Marshfield Clinic, Marshfield, Wisconsin
  - St. Joseph's Hospital, Milwaukee, Wisconsin
  - Waukesha Memorial Hospital, Inc, Waukesha, Wisconsin
  - Children's Corporate Center, Wauwatosa, Wisconsin
- Argentina (4):
  - Hospital Peiade Interzonal General de Augodos, Buenos Aires
  - Hospital General De Ninos Pedro De Elizalde, Buenos Aires
  - Sanatorio Trinidad, Capital Federal
  - Hospital Materno Neonatal, Córdoba
- Australia (10):
  - The Canberra Hospital, Garran, Australian Capital Territory
  - John Hunter Children's Hospital, New Lambton, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Children's Hospital (Brisbane), Herston, Queensland
  - Peninsula Clinical Research Centre, Kippa-Ring, Queensland
  - Mater Mothers Hospital Raymond Terrace, South Brisbane, Queensland
  - Royal Hobart Hospital, Hobart, Tasmania
  - Royal Children's Hospital (Melbourne), Parkville, Victoria
  - Princess Margaret Children's Hospital, Subiaco, Western Australia
  - Women's and Children's Hospital, North Adelaide
- Austria (4):
  - Universitatsklinik fur Kinder und Jugenheilkunde, Graz, Graz
  - LandesKrankenHaus Tulln, Kinderabteilung, Tulln
  - Allgemeines KrankenHaus Universitatsklinkiken Wein, Vienna
  - SMZ-Ost Donauspital Wien, Vienna
- Brazil (8):
  - Hospital e Maternidade Celso Pierro-Puccamp, Campinas
  - Mernidade Nossa Senhora De Fatima, Curitiba
  - Hospital De Clinicas Da UFPR, Curitiba
  - Hospital Sao Lucas da PUC-RS de Riberiao Perto da Universidade de Sao Paulo, Porto Alegre
  - Hospital Das Clinicas Da Faculdade De Medicina, Ribeirão Preto
  - Santa Casa de Misericordia de Sao Paulo, São Paulo
  - Hospital e Maternidade Santa Marina, São Paulo
  - Hospital Universitario de Universidade de Sao Paulo, São Paulo
- Bulgaria (9):
  - Multifunctional Hospital for Active Treatment "Pleven", Pleven
  - University Multifunctional Hospital for Active Treatment "St. George" Neonatology Clinic, Plovdiv
  - University Multifunctional Hospital for Active Treatment "St. George" Clinic of Pediatrics, Plovdiv
  - Multifunctional Hospital for Active Treatment - Plovdiv, Plovdiv
  - Regional Hospital of Pulmonary Diseases, Rousse
  - Specialized Hospital for Active Treatment of Cardio-vascular Diseases, Sofia
  - Specialized Hospital for Active Treatment of Obstetrics and Gynaecology"-"Maichin Dom", Sofia
  - Specialized Hospital for Active Treatment of Pediatric Diseases, Sofia
  - Multifunctional Hospital for Active Treatment "St. Marina", Varna
- Canada (14):
  - Alberta Children's Hospital, Calgary
  - Queen Elizabeth Hospital, Charlottetown
  - University Of Alberta/Stollery Children's Hospital, Edmonton
  - Dalhousie University IWK Health Centre, Halifax
  - Mcmaster Children's Hospital, Hamilton
  - McGill University Health Centre Monteal Children's Hospital, Montreal
  - Sainte Justine Hospital, Montreal
  - Children's Hospital of Eastern Ontario, Ottawa
  - Centre Hospitalier de L'Universite Laval, Québec
  - Royal University Hospital, Saskatoon
  - Children's And Women's Hospital of BC, Vancouver
  - Victoria General Hospital, Victoria
  - Windsor Regional Hospital, Windsor
  - Manitoba Institute Of Child Health University of Manitoba, Winnipeg
- Chile (6):
  - Hospital San Jose, Independencia
  - Hospital Clinico de la Universidad de Chile, Independencia
  - Hospital Dr. Sotero Del Rio, Puente Alto
  - Hospital Dr. Feliz Buines Cerda, Quinta Normal
  - Hospital Clinico San Borja Arriaran, Santiago
  - Hospital Padre Hurtado, Santiago
- Czechia (12):
  - Nemocnice CB, České Budějovice
  - FN Hradec Kralove Detska klinika, Hradec Králové
  - Nemocnice s poliklinikou v Moste, Most
  - Fakultni nemocnice, Olomouc
  - FNsP Ostrava, Ostrava
  - FN Plzen, Plzen-Bory
  - FN Plzen, Plzen-Lochotin
  - Vfn 1.Lf Uk, Prague
  - Fakultni Thomayerova nemocnice S poliklinkou, Prague
  - Ustav pro peci o matku a dite, Prague
  - FN Motol Novorozenecke oddeleni, Prague
  - Batova krajska nemocnice Zlin, Zlín
- Denmark (4):
  - Paediatrisk Afdeling Herning Centralsygehus, Herning
  - Hillerod Sygehus Helsevej 2, Hillerød
  - Hvidovre Hospital, Hvidovre
  - Sygehus Viborg, Viborg
- France (16):
  - Service de Medecine Neonatale et de reanimation pediatrique, Amiens
  - CHU Angers, Angers
  - CHU de Besancon-Hopital Saint-Jacques, Besançon
  - CHU Bordeaux/Hopital des enfants/Unite de Neonatologie B, Bordeaux
  - CH Chambery, Chambéry
  - CHU Dijon, Dijon
  - Hopital Jeanne de Flandre, Lille
  - CHU Nord, Marseille
  - CHU Montpellier/Hoptial Arnaud de Villeneuve, Montpellier
  - CHU de Nantes/Hospital Mere-Enfant, Nantes
  - CHI Poissy/St Germain en Laye, Poissy
  - CHU Rennes/Hopital Sud, Rennes
  - CHU Rouen, Rouen
  - CH Pierre Haute, Strasbourg
  - CHU Toulouse-Hopital des Enfants, Toulouse
  - Centre Pediatrique Gatien de Clocheville, Tours
- Germany (17):
  - Ruhr-Uni St. Josef Hospital, Bochum
  - Klinikum Duisburg, Wedau Kliniken, Duisburg
  - Uni-Kinderklinik, Düsseldorf
  - Klinik fur Kinder und Jugendliche, Erlangen
  - Zentrum Klinische Studien/Universtatsklinikum Freiburg, Freiburg im Breisgau
  - Universtatsklinikum Gottingen, Göttingen
  - Wittenberg/Zentrum: fur Kinderheilkunde, Universitatsklinik und Poliklinik fur Kinder and Jugendmedizin, Halle
  - Stiftung Hannoversche, Hanover
  - Im Neuenheimer Feld 153, Heidelberg
  - Klinik und Poliklinik und Jugendiche der Universitat Leipzig, Leipzig
  - Universitatskinderlinik/Zentrum Fur klinische Studien, Mainz
  - Kinderklinik und Kinderpoliklinik, München
  - Stadtisches Krankenhaus Muchen-Harlaching, München
  - Evangelischisches Krankenhaus, Oberhausen
  - Klinikum Oldenberg, Oldenberg
  - Klinikum Rosenheim, Rosenheim
  - Asklepios Kinderklinik Sankt Augustin GmbH, Sankt Augustin
- Greece (5):
  - "P&A Kyriakou" Children's hospital, Athens
  - Aghia Sofia Children hospital, Athens
  - Aristotele University of Thessaloniki, General "AXEPA" Hospital, Thessaloniki
  - Hippokration Hospital, University of Thessaloniki, Thessaloniki
  - General hospital "Papageorgiou", Thessaloniki
- Hungary (11):
  - Semmelweis Univ., Budapest
  - Semmelweis University, Budapest
  - Schopf-Merei Agost Hospital, Budapest
  - DEOEC Neonatology Division, Debrecen
  - DEOEC, Dept. of Pediatry, Debrecen
  - Petz Aladar Teaching Hospital, Győr
  - Borsod-Abaúj-Zemplén Megyei Önkormányzat Kórháza, Miskolc
  - Josa Andras Hospital, Nyíregyháza
  - University of Pecs, Pécs
  - Univ. of Pecs, Pécs
  - Csolnoky Ferenc Hospital, Veszprém
- Children's hospital, Landspitali University Hospital, Reykjavik, Iceland
- Israel (16):
  - HaEmek Medical Center, Afula
  - Barzilai Medical Center, Ashkelon
  - Soroka Medical Center, Beersheba
  - Bnei Zion Medical Center, Haifa
  - Rambam Medical Center, Haifa
  - Carmel Medical Center, Haifa
  - Wolfson Medical Center, Holon
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Ein-Kerem Medical Center, Jerusalem
  - Sapir Medical Center, Kfar Saba
  - Laniado Medical Center, Netanya
  - Schneider Medical Center, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - Sourasky Medical Center (Ichilov), Tel Aviv
  - Chaim Sheba Medical Center, Tel Litwinsky
  - Poria Medical Center, Tiberias
- Italy (15):
  - Presio Ospedaliero di Alta Specializzazione "G. Salesi" - Azienda Ospedaliera Universitaria - Ospedali Riuniti "Umberto I - G.M. Lancisi - G. Salesi", Ancona
  - Ospedali Riuniti di Bergamo - Azienda Ospedaliera/Unità Operativa di Patologia Neonatale, Bergamo
  - Azienda Ospedaliera di Bologna - Policlinico S. Orsola - Malpighi, Bologna
  - Ospedale Generale di Bolzano, Bolzano
  - Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliera S. Croce e Carle, Cuneo
  - Azienda Ospedaliera Universitaria, Foggia
  - Azienda USL di Imola - Ospedale di Imola, Imola
  - Ospedale Alessandro Manzoni Lecco - Presidio dell'Azienda Ospedaliera "Ospedale di Lecco", Lecco
  - Azienda Ospedaliera Universitaria Policlinico Gaetano Martino, Messina
  - Azienda Ospedaliera San Gerardo, Monza
  - Azienda Ospedaliera di Parma, Parma
  - Azienda Ospedaliera Universitaria Pisana - Ospedale S. Chiara, Pisa
  - Azienda Sanitaria Ospedaliera O.I.R.M.-S. Anna, Torino
  - Azienda Ospedaliera S. Maria della Misericordoa Struttura Operativa Complessa di Patologia Neonatale e terapia Intesiva Neonatale, Udine
- New Zealand (4):
  - Middlemore Hospital, Auckland
  - Dunedin Hospital, Dunedin
  - Waikato Hospital, Hamilton
  - Palmerston North Hospital, Palmerston North
- Poland (15):
  - Klinika Neonatologii AM w Białymstoku, Bialystok
  - Samodzielny Publiczny Zakład Opieki Zdrowotnej Wojewódzki Szpital im. dr Jana Biziela w Bydgoszczy, Oddział Noworodków, Wcześniaków I Intensywnej Terapii Noworodka, Bydgoszcz
  - Oddział Pediatrii i Kardiologii z pododdziałem Patologii Noworodka, Bydgoszcz
  - Wojewódzki Szpital Specjalistyczny, Oddział Dziecięcy, Częstochowa
  - Samodzielny Publiczny Szpital Kliniczny nr 1, Klinika Neonatologii, Gdansk
  - Szpital Morski im. PCK, Oddział Dziecięcy, Gdynia
  - Oddzial Kliniczny Kliniki Neonatologii Szpitala Uniwersyteckiego w Krakowie, Krakow
  - Szpital Kliniczny nr 4 im.M.Konopnickiej, Oddział Intensywnej Terapii i Anestezjologii, Lodz
  - Klinika Neonatologii, Instytut Centrum Zdrowia Matki Polki, Lodz
  - Dziecięcy Szpital Kliniczny im. Prof. dr hab. n. med. Antoniego Gębali w Lublinie, Lublin
  - Katedra i Klinika Neonatologii AM w Poznaniu, Poznan
  - II Klinika Chorób Dzieci PAM, Samodzielny Publiczny, Szczecin
  - Klinika Neonatologii AM w Warszawie, Warsaw
  - Klinika Niemowlęca, Instytut Pomnik - Centrum Zdrowia Dziecka, Warsaw
  - Niepubliczny Zakład Opieki Zdrowotnej Salmed s.c., Łęczna
- Russia (7):
  - Pediatric City Hospital #13, Moscow
  - Morozovsky Pediatric City Hospital, Moscow
  - St. Petersburg City Outpatient Hospital #45, Saint Petersburg
  - Saint-Petersburg State Pediatric Medical Academy, Saint Petersburg
  - St. Petersburg State Pediatric Medical Academy, Saint Petersburg
  - Pediatric City Hospital #1, Saint Petersburg
  - Smolensk State Medical Academy, Smolensk
- Spain (25):
  - Hospital Juan Canalejo, A Coruña
  - Hospital Clinic y Maternistat - Barcelona, Barcelona
  - Hospital Sant Joan de Déu (Barcelona), Barcelona
  - Hospital Reina Sofia, Córdoba
  - Hospital de Cruces, Cruces
  - Hospital Josep Trueta, Girona
  - Hospital Virgen de las Nieves, Granada
  - Hospital de Donostia (San Sebastian), Guipuzcoa
  - Hospital Materno Infantil deJaén, Jaén
  - Hospital General de Jerez, Jerez de la Frontera
  - Hospital Materno Infantil de Canarias, Las Palmas de Gran Canaria
  - Hospital Clínico San Carlos, Madrid
  - Hospital La Paz- Madrid, Madrid
  - Hospital Severo Ochoa, Madrid
  - Hospital Materno Infantil/Neumología pediátrica, Málaga
  - Hospital Central de Asturias, Oviedo
  - Hospital Clinico de Salamanca, Salamanca
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela
  - Hospital Maternal Virgen del Rocío, Seville
  - Hospital Virgen Macarena, Seville
  - Hospital Joan XXIII, Tarragona
  - Hospital Universitario La Fe Maternidad, Valencia
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Xeral-Cíes, Vigo
- Sweden (5):
  - Mälarsjukhuset, Eskilstuna
  - The Queen Silvia Children's Hospital, Gothenburg
  - Karolinska University Hospital Solna, Stockholm
  - Danderyds Sjukhus, Stockholm
  - Uppsala University Hospital, Uppsala
- Turkey (Türkiye) (4):
  - Hacettepe Üniversitesi İhsan Doğramacı Çocuk Hastanesi Neonatoloji Ünitesi, Ankara
  - Ankara Üniversitesi, Ankara
  - Ege Üniversitesi Tıp Fakültesi, Izmir
  - Dokuz Eylül Üniversitesi Tıp Fakültesi, Izmir
- United Kingdom (11):
  - Birmingham Heartlands Hospital, Birmingham
  - Dumfries and Galloway Royal Infirmary, Dumfries
  - Children's Respiratory Medicine Division of Maternal and Child Health Sciences Ninewells Hospital, Dundee
  - Medway Maritime Hospital, Gillingham Kent
  - Princess Anne Hospital, Hants
  - Claredon Wing, Leeds General Infirmary, Leeds
  - St James' University Hospital, Leeds
  - James Cook University Hospital, Middlesbrough
  - Queen's Medical Centre Nottingham University Hospital, Nottingham
  - Sheffield Children's Hospital, Sheffield
  - Royal Hampshire County Hospital, Winchester

REFERENCES:
- [Result] Carbonell-Estrany X, Simoes EA, Dagan R, Hall CB, Harris B, Hultquist M, Connor EM, Losonsky GA; Motavizumab Study Group. Motavizumab for prophylaxis of respiratory syncytial virus in high-risk children: a noninferiority trial. Pediatrics. 2010 Jan;125(1):e35-51. doi: 10.1542/peds.2008-1036. Epub 2009 Dec 14. PMID 20008423

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 6,635 children were randomized in a 1:1 ratio at 347 centers in 24 countries within the Northern and Southern hemispheres between 01/Nov/2004 and 09/Dec/2005; each child participated in the study for a single RSV season.
Pre-assignment Details: Randomization was blocked by study site and stratified according to presence/absence of CLD of prematurity requiring medical intervention/management.
Groups:
- Motavizumab: Motavizumab, 15 mg/kg administered intramuscularly for 5 monthly doses
Period: Overall Study
Arm/Group | Palivizumab | Motavizumab
Started | 3306 | 3329
Completed | 3246 | 3270
Not Completed | 60 | 59
Not completed — Death | 3 | 8
Not completed — Withdrawal of consent | 31 | 30
Not completed — Lost to Follow-up | 26 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Palivizumab | Motavizumab | Total
Number analyzed (Participants) | 3306 | 3329 | 6635
Age Continuous [Mean (Standard Deviation); unit: months] | 3.98 (3.78) | 3.99 (3.75) | 3.99 (3.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1495 | 1513 | 3008
  Male | 1811 | 1816 | 3627
Region of Enrollment [Number; unit: participants]
  United States | 1130 | 1167 | 2297
  Greece | 32 | 34 | 66
  Spain | 191 | 181 | 372
  Turkey | 36 | 42 | 78
  Austria | 35 | 34 | 69
  Russian Federation | 42 | 45 | 87
  Israel | 301 | 305 | 606
  Chile | 93 | 87 | 180
  United Kingdom | 89 | 90 | 179
  Italy | 93 | 96 | 189
  France | 107 | 111 | 218
  Hungary | 198 | 192 | 390
  Czech Republic | 171 | 177 | 348
  Canada | 134 | 132 | 266
  Argentina | 38 | 34 | 72
  Poland | 106 | 105 | 211
  Brazil | 69 | 66 | 135
  Australia | 85 | 81 | 166
  Denmark | 30 | 27 | 57
  Bulgaria | 95 | 101 | 196
  Iceland | 20 | 19 | 39
  Germany | 131 | 122 | 253
  New Zealand | 26 | 26 | 52
  Sweden | 54 | 55 | 109

OUTCOME MEASURES:

1. Primary Outcome: Incidence of RSV Hospitalization (Includes Deaths by RSV)
Description: RSV hospitalization was defined as 1) a respiratory hospitalization with a positive RSV test (primary), 2) a new onset of lower respiratory symptoms in an already hospitalized child, with an objective measure of worsening respiratory status and positive RSV test (nosocomial), or 3) death demonstrated to have been caused by RSV (by autopsy or clinical history and virologic evidence).
Time Frame: Days 0 - 150
Population: The Intent-to-Treat (ITT) Population included all patients randomized into the study.
Measure: Number; unit: Participants
Arm/Group | Palivizumab | Motavizumab
Number analyzed (Participants) | 3306 | 3329
Participants | 62 | 46
Statistical Analysis 1: Comparison: Palivizumab vs Motavizumab; ITT population; Test type: Non-Inferiority or Equivalence — Confidence interval and relative risk adjusted for the stratification factor of presence or absence of CLD of prematurity as specified on the CRF; t-test, 2 sided; Risk Ratio (RR) = 0.740, 95% CI 2-sided [0.503 to 1.083] — Relative risk was calculated as (Pn/Ps) where Pn is the proportion of patients with RSV hospitalization in the motavizumab group and Ps is the proportion of patients with RSV hospitalization in the palivizumab group

2. Primary Outcome: Number of Participants Reporting Any Adverse Events (AEs)
Description: Number of participants reporting one or more AEs
Time Frame: Days 0 - 150
Population: The Safety Population included all patients who received any study drug and had any safety follow-up.
Measure: Number; unit: participants
Arm/Group | Palivizumab | Motavizumab
Number analyzed (Participants) | 3298 | 3315
participants | 2837 | 2839

3. Primary Outcome: Number of Participants Reporting Any Related AEs
Description: Number of participants reporting one or more AEs considered related to study drug by the investigator
Time Frame: Days 0 - 150
Population: The Safety Population included all patients who received any study drug and had any safety follow-up.
Measure: Number; unit: participants
Arm/Group | Palivizumab | Motavizumab
Number analyzed (Participants) | 3298 | 3315
participants | 258 | 298

4. Primary Outcome: Number of Participants Reporting Any Serious Adverse Events (SAEs)
Description: Number of participants reporting one or more SAEs
Time Frame: Days 0 - 150
Population: The Safety Population included all patients who received any study drug and had any safety follow-up.
Measure: Number; unit: participants
Arm/Group | Palivizumab | Motavizumab
Number analyzed (Participants) | 3298 | 3315
participants | 506 | 485

5. Primary Outcome: Number of Participants Reporting Any Related SAEs
Description: Number of participants reporting one or more SAEs considered related to study drug by the investigator
Time Frame: Days 0 - 150
Population: The Safety Population included all patients who received any study drug and had any safety follow-up.
Measure: Number; unit: participants
Arm/Group | Palivizumab | Motavizumab
Number analyzed (Participants) | 3298 | 3315
participants | 8 | 9

6. Primary Outcome: Number of Participants Reporting AEs by Highest Severity Grade
Description: Adverse events events were graded by severity; Level 1, 2, 3, or 4
Time Frame: Days 0 - 150
Population: The Safety Population included all patients who received any study drug and had any safety follow-up.
Measure: Number; unit: participants
Arm/Group | Palivizumab | Motavizumab
Number analyzed (Participants) | 3298 | 3315
participants
  Level 1 | 1478 | 1538
  Level 2 | 1006 | 976
  Level 3 | 292 | 271
  Level 4 | 61 | 54

7. Primary Outcome: Number of Participants Who Discontinued Study Drug Due to AEs
Time Frame: Days 0 - 150
Population: The Safety Population included all patients who received any study drug and had any safety follow-up.
Measure: Number; unit: participants
Arm/Group | Palivizumab | Motavizumab
Number analyzed (Participants) | 3298 | 3315
participants | 10 | 13

8. Primary Outcome: Number of Participants Who Died
Time Frame: Days 0 - 150
Population: The Safety Population included all patients who received any study drug and had any safety follow-up.
Measure: Number; unit: participants
Arm/Group | Palivizumab | Motavizumab
Number analyzed (Participants) | 3298 | 3315
participants | 4 | 8

9. Primary Outcome: Number of Participants Reporting Changes in Vital Signs From Baseline
Description: Vital signs that were in a higher toxicity grade than observed at baseline were to be recorded as AEs
Time Frame: Days 0 - 150
Population: The Safety Population included all patients who received any study drug and had any safety follow-up.
Measure: Number; unit: participants
Arm/Group | Palivizumab | Motavizumab
Number analyzed (Participants) | 3298 | 3315
participants
  Fever neonatal | 0 | 2
  Hyperpyrexia | 0 | 1
  Hyperthermia | 3 | 3
  Hypothermia | 2 | 2
  Pyrexia | 559 | 544
  Hypertension | 4 | 4
  Hypotension | 2 | 2
  Arrhythmia | 1 | 0
  Bradycardia | 10 | 4
  Tachycardia | 4 | 6

10. Secondary Outcome: The Incidence of Outpatient Medically-attended Lower Respiratory Illness (LRI)
Description: LRI was defined as an event of bronchiolitis or pneumonia or the occurance of a lower tract infectious illness as determined by the PI based on medical history, signs, and symptoms.
Time Frame: Day 0 - 150
Population: The Intent-to-Treat (ITT) Population included all patients randomized into the study.
Measure: Number; unit: Participant
Arm/Group | Palivizumab | Motavizumab
Number analyzed (Participants) | 3306 | 3329
Participant | 696 | 648
Statistical Analysis 1: Comparison: Palivizumab vs Motavizumab; Test type: Non-Inferiority or Equivalence — A CMH approach stratified by presence or absence of CLD of prematurity requiring medical intervention was used; p = 0.110, Cochran-Mantel-Haenszel — Test stratified by presence or absence of CLD of prematurity specified on the CRF

11. Secondary Outcome: The Incidence of RSV-specific Medically-attended Outpatient Lower Respiratory Illnesses (LRIs) Between Treatment Groups
Description: The RSV-specific LRI was defined as an outpatient medically-attended LRI associated with a positive RSV test and was not inclusive of events that required hospitalization.
Time Frame: Days 0 - 150
Population: Subjects were from a pre-specified subsets of sites participating in the nasal secretion sample collection for this endpoint.
Measure: Number; unit: Participants
Arm/Group | Palivizumab | Motavizumab
Number analyzed (Participants) | 1183 | 1227
Participants | 46 | 24
Statistical Analysis 1: Comparison: Palivizumab vs Motavizumab; Test type: Non-Inferiority or Equivalence — A CMH approach stratified by presence or absence of CLD of prematurity requiring medical intervention was used; p = 0.005, Cochran-Mantel-Haenszel — No adjustment for multiple comparisons; The CMH test was stratified by presence or absence of CLD of prematurity as specified on the CRF

12. Secondary Outcome: The Incidence of Medically-attended Otitis Media (OM) Infections
Description: Otitis media (OM) was to be recorded as the diagnosis if the following terms were used by the medical care provider: acute OM, acute tympanic membrane (TM) perforation, bulging TM, red TM with fever, OM with effusion, or middle ear effusion. A new episode was defined as a physician-diagnosed OM in either ear after a normal middle ear exam of the ear in question or an episode of acute OM greater than or equal to 21 days after resolution of the previous episode. A diagnosis of persistent middle ear effusion was not to be recorded as a new OM event.
Time Frame: Days 0 - 150
Population: The Intent-to-Treat (ITT) Population included all patients randomized into the study.
Measure: Number; unit: Participants
Arm/Group | Palivizumab | Motavizumab
Number analyzed (Participants) | 3306 | 3329
Participants
  Overall incidence | 461 | 484
  0 infections | 2845 | 2845
  1 infection | 329 | 360
  2 infections | 100 | 91
  3 or more infections | 32 | 33
Statistical Analysis 1: Comparison: Palivizumab vs Motavizumab; P-value is for overall incidence; Test type: Non-Inferiority or Equivalence — A CMH approach stratified by presence or absence of CLD of prematurity requiring medical intervention was used; p = 0.476, Van Eleteren test; Test stratified by presence or absence of CLD of prematurity specified on the CRF

13. Secondary Outcome: The Frequency of Prescribed Antibiotics for Medically-attended LRI
Description: The average number of presciptions per event per subject was summarized for each treatment group.
Time Frame: Days 0 - 150
Population: The Intent-to-Treat (ITT) Population included all patients randomized into the study.
Measure: Mean (Standard Deviation); unit: Number of prescriptions
Arm/Group | Palivizumab | Motavizumab
Number analyzed (Participants) | 3306 | 3329
Number of prescriptions | 0.32 (0.02) | 0.30 (0.02)
Statistical Analysis 1: Comparison: Palivizumab vs Motavizumab; Test type: Non-Inferiority or Equivalence — A CMH approach stratified by presence or absence of CLD of prematurity requiring medical intervention was used; p = 0.493, Van Eleteren test — Test stratified by presence or absence of CLD of prematurity specified on the CRF

14. Secondary Outcome: The Frequency of Prescribed Antibiotics for Medically-attended OM Infections
Description: The average number of presciptions per event per subject was summarized for each treatment group.
Time Frame: Days 0 - 150
Population: The Intent-to-Treat (ITT) Population included all patients randomized into the study.
Measure: Mean (Standard Deviation); unit: number of prescriptions
Arm/Group | Palivizumab | Motavizumab
Number analyzed (Participants) | 3306 | 3329
number of prescriptions | 1.08 (0.003) | 1.10 (0.003)
Statistical Analysis 1: Comparison: Palivizumab vs Motavizumab; Test type: Non-Inferiority or Equivalence — A CMH approach stratified by presence or absence of CLD of prematurity requiring medical intervention was used; p = 0.652, Van Eleteren test — Test stratified by presence or absence of CLD of prematurity specified on the CRF

15. Secondary Outcome: The Number of Participants With Anti-motavizumab Antibodies
Description: Detection of anti-motavizumab antibodies was defined as a titer with a dilution value equal to or greater than 1:10.
Time Frame: Day 0 - 120
Population: N varied at different timepoints: at pre-dose 1 N=3193; at 30 days post-dose 1 N=998; at 30 days post-dose 2 N=1049; at 30 days post-dose 3 N=1049; at 30 days post-dose 4, N=3013; at any time post baseline, N=3217
Measure: Number; unit: participants
Arm/Group | Motavizumab
Number analyzed (Participants) | 3217
participants
  Pre-dose 1 | 7
  30 Days Post-Dose 1 | 1
  30 Days Post-Dose 2 | 1
  30 Days Post-Dose 3 | 7
  30 Days Post-Dose 4 | 18
  At any time post baseline | 22

16. Secondary Outcome: The Serum Concentrations of Motavizumab at Day 0
Description: Mean serum concentrations of motavizumab at Day 0
Time Frame: Day 0
Population: The Pharmacokinetics/Immunogenicity (PK/IM) Population included all patients who received study drug and who did not receive non-study commercial palivizumab within 3 months prior to receiving the first dose of study drug.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Motavizumab
Number analyzed (Participants) | 3147
ug/mL | 0.01193 (0.2072)

17. Secondary Outcome: The Trough Serum Concentrations of Motavizumab at 30 Days Post Dose 1
Description: Mean serum concentrations of motavizumab at 30 days post Dose 1
Time Frame: 30 days post Dose 1
Population: The Pharmacokinetics/Immunogenicity (PK/IM) Population included all patients who received study drug and who did not receive non-study commercial palivizumab within 3 months prior to receiving the first dose of study drug. Includes subjects with both baseline and a post-dose 1 measurements
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Motavizumab
Number analyzed (Participants) | 974
ug/mL | 45.95 (15.17)

18. Secondary Outcome: The Trough Serum Concentrations of Motavizumab at 30 Days Post Dose 2
Description: Mean serum concentrations of motavizumab at 30 days post Dose 2
Time Frame: 30 days post Dose 2
Population: The Pharmacokinetics/Immunogenicity (PK/IM) Population included all patients who received study drug and who did not receive non-study commercial palivizumab within 3 months prior to receiving the first dose of study drug. Includes subjects with both baseline and a post-dose 2 measurements
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Motavizumab
Number analyzed (Participants) | 915
ug/mL | 64.59 (25.60)

19. Secondary Outcome: The Trough Serum Concentrations of Motavizumab at 30 Days Post Dose 3
Description: Mean serum concentrations of motavizumab at 30 days post Dose 3
Time Frame: 30 days post Dose 3
Population: The Pharmacokinetics/Immunogenicity (PK/IM) Population included all patients who received study drug and who did not receive non-study commercial palivizumab within 3 months prior to receiving the first dose of study drug. Includes subjects with both baseline and a post-dose 3 measurements
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Motavizumab
Number analyzed (Participants) | 918
ug/mL | 80.24 (31.22)

20. Secondary Outcome: The Trough Serum Concentrations of Motavizumab at 30 Days Post Dose 4
Description: Mean serum concentrations of motavizumab at 30 days post Dose 4
Time Frame: 30 days post Dose 4
Population: The Pharmacokinetics/Immunogenicity (PK/IM) Population included all patients who received study drug and who did not receive non-study commercial palivizumab within 3 months prior to receiving the first dose of study drug. Includes subjects with both baseline and a post-dose 4 measurements
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Motavizumab
Number analyzed (Participants) | 2669
ug/mL | 88.52 (35.43)

ADVERSE EVENTS:
Time Frame: Day 0 - Day 150
Arm/Group | Palivizumab | Motavizumab
Serious Adverse Events (participants affected / at risk) | 506/3298 | 485/3315
Other Adverse Events (participants affected / at risk) | 2777/3298 | 2784/3315
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Palivizumab (N=3298) | Motavizumab (N=3315)
ANAEMIA (Blood and lymphatic system disorders) | 4 (4) | 5 (5)
ANAEMIA NEONATAL (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
CYCLIC NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
HAEMOLYTIC URAEMIC SYNDROME (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
ATRIAL THROMBOSIS (Cardiac disorders) | 0 (0) | 1 (1)
BRADYCARDIA (Cardiac disorders) | 4 (4) | 2 (2)
CARDIAC ARREST (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC FAILURE HIGH OUTPUT (Cardiac disorders) | 1 (1) | 0 (0)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 (1) | 0 (0)
CARDIOGENIC SHOCK (Cardiac disorders) | 1 (1) | 0 (0)
CYANOSIS (Cardiac disorders) | 2 (2) | 1 (1)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1)
ACRODERMATITIS ENTEROPATHICA (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
ANAL ATRESIA (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
ANKYLOGLOSSIA CONGENITAL (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
BRANCHIAL CLEFT CYST (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
CEREBRAL PALSY (Congenital, familial and genetic disorders) | 1 (2) | 0 (0)
CLEFT LIP (Congenital, familial and genetic disorders) | 0 (0) | 2 (2)
CLEFT LIP AND PALATE (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
CLEFT PALATE (Congenital, familial and genetic disorders) | 2 (2) | 0 (0)
DACRYOSTENOSIS CONGENITAL (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
DERMOID CYST (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
HAMARTOMA (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
HIP DYSPLASIA (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
LIMB REDUCTION DEFECT (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
PHIMOSIS (Congenital, familial and genetic disorders) | 1 (1) | 1 (1)
PILONIDAL CYST CONGENITAL (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
PYLORIC STENOSIS (Congenital, familial and genetic disorders) | 1 (1) | 1 (1)
RESPIRATORY TRACT MALFORMATION (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
SYNDACTYLY (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
TALIPES (Congenital, familial and genetic disorders) | 2 (2) | 2 (7)
TRACHEO-OESOPHAGEAL FISTULA (Congenital, familial and genetic disorders) | 1 (3) | 0 (0)
VENTRICULAR SEPTAL DEFECT (Congenital, familial and genetic disorders) | 1 (2) | 0 (0)
DEAFNESS (Ear and labyrinth disorders) | 0 (0) | 1 (1)
PAPILLOEDEMA (Eye disorders) | 0 (0) | 1 (1)
RETINOPATHY OF PREMATURITY (Eye disorders) | 7 (7) | 5 (5)
RETINOPATHY PROLIFERATIVE (Eye disorders) | 0 (0) | 1 (1)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 (3) | 2 (2)
ABDOMINAL STRANGULATED HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
ANAL FISTULA (Gastrointestinal disorders) | 1 (1) | 0 (0)
COLONIC STENOSIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 2 (2)
DIARRHOEA (Gastrointestinal disorders) | 5 (6) | 2 (2)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 1 (1)
DYSPHAGIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
ENTERITIS (Gastrointestinal disorders) | 1 (1) | 1 (1)
ENTEROCOLITIS (Gastrointestinal disorders) | 1 (1) | 2 (2)
ENTEROCUTANEOUS FISTULA (Gastrointestinal disorders) | 1 (1) | 0 (0)
FAECES DISCOLOURED (Gastrointestinal disorders) | 0 (0) | 1 (1)
FLATULENCE (Gastrointestinal disorders) | 2 (2) | 0 (0)
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (2)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 21 (22) | 18 (20)
HIATUS HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
ILEUS (Gastrointestinal disorders) | 0 (0) | 1 (1)
INGUINAL HERNIA (Gastrointestinal disorders) | 57 (58) | 56 (58)
INGUINAL HERNIA, OBSTRUCTIVE (Gastrointestinal disorders) | 3 (4) | 1 (1)
INTUSSUSCEPTION (Gastrointestinal disorders) | 1 (1) | 0 (0)
NECROTISING COLITIS (Gastrointestinal disorders) | 1 (1) | 2 (2)
OESOPHAGEAL MASS (Gastrointestinal disorders) | 0 (0) | 1 (1)
PANCREATITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
REFLUX OESOPHAGITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
REGURGITATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
UMBILICAL HERNIA (Gastrointestinal disorders) | 1 (1) | 1 (1)
VOMITING (Gastrointestinal disorders) | 3 (3) | 5 (5)
FEVER NEONATAL (General disorders) | 0 (0) | 2 (2)
HERNIA (General disorders) | 1 (1) | 0 (0)
HERNIA OBSTRUCTIVE (General disorders) | 0 (0) | 1 (1)
HYPOTHERMIA (General disorders) | 1 (1) | 1 (1)
MALAISE (General disorders) | 0 (0) | 1 (1)
OEDEMA PERIPHERAL (General disorders) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 9 (9) | 10 (11)
SUDDEN DEATH (General disorders) | 0 (0) | 1 (1)
SUDDEN INFANT DEATH SYNDROME (General disorders) | 2 (2) | 3 (3)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
CHOLESTASIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
HEPATIC CYST (Hepatobiliary disorders) | 1 (1) | 0 (0)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 1 (1) | 1 (1)
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 1 (1)
HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 1 (1)
IMMUNISATION REACTION (Immune system disorders) | 1 (1) | 0 (0)
ABSCESS LIMB (Infections and infestations) | 0 (0) | 1 (1)
ABSCESS NECK (Infections and infestations) | 1 (1) | 0 (0)
ADENOVIRAL UPPER RESPIRATORY INFECTION (Infections and infestations) | 0 (0) | 1 (1)
BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1)
BACTERIAL ABSCESS CENTRAL NERVOUS SYSTEM (Infections and infestations) | 0 (0) | 1 (1)
BACTERIAL PYELONEPHRITIS (Infections and infestations) | 0 (0) | 1 (1)
BACTERIAL TRACHEITIS (Infections and infestations) | 1 (2) | 0 (0)
BRONCHIOLITIS (Infections and infestations) | 78 (88) | 71 (87)
BRONCHITIS (Infections and infestations) | 36 (46) | 35 (39)
BRONCHITIS VIRAL (Infections and infestations) | 3 (3) | 0 (0)
BRONCHOPNEUMONIA (Infections and infestations) | 8 (8) | 12 (13)
CATHETER SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
CELLULITIS (Infections and infestations) | 3 (3) | 1 (1)
CENTRAL LINE INFECTION (Infections and infestations) | 0 (0) | 1 (1)
CLOSTRIDIAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
CROUP INFECTIOUS (Infections and infestations) | 7 (8) | 6 (6)
CYTOMEGALOVIRUS INFECTION (Infections and infestations) | 0 (0) | 1 (1)
DACRYOCYSTITIS (Infections and infestations) | 1 (1) | 1 (1)
DYSENTERY (Infections and infestations) | 1 (1) | 0 (0)
ENTEROBACTER BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1)
ENTEROCOLITIS VIRAL (Infections and infestations) | 0 (0) | 1 (1)
ESCHERICHIA SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 2 (2) | 0 (0)
EXANTHEMA SUBITUM (Infections and infestations) | 1 (1) | 0 (0)
EXTERNAL EAR CELLULITIS (Infections and infestations) | 0 (0) | 1 (1)
GASTROENTERITIS (Infections and infestations) | 31 (31) | 27 (28)
GASTROENTERITIS ADENOVIRUS (Infections and infestations) | 1 (1) | 0 (0)
GASTROENTERITIS ESCHERICHIA COLI (Infections and infestations) | 1 (1) | 0 (0)
GASTROENTERITIS ROTAVIRUS (Infections and infestations) | 21 (21) | 13 (15)
GASTROENTERITIS SALMONELLA (Infections and infestations) | 0 (0) | 1 (1)
GASTROENTERITIS VIRAL (Infections and infestations) | 6 (6) | 2 (2)
HERPES ZOSTER (Infections and infestations) | 1 (1) | 0 (0)
IMPETIGO (Infections and infestations) | 1 (1) | 0 (0)
INFECTION (Infections and infestations) | 1 (1) | 0 (0)
INFLUENZA (Infections and infestations) | 3 (3) | 4 (4)
LARYNGITIS (Infections and infestations) | 5 (7) | 5 (5)
LOBAR PNEUMONIA (Infections and infestations) | 3 (3) | 2 (2)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 8 (8) | 6 (6)
LOWER RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 1 (1) | 0 (0)
LUNG ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
LYMPHADENITIS BACTERIAL (Infections and infestations) | 1 (1) | 1 (1)
MENINGITIS VIRAL (Infections and infestations) | 0 (0) | 1 (1)
NASOPHARYNGITIS (Infections and infestations) | 3 (3) | 2 (2)
ORAL CANDIDIASIS (Infections and infestations) | 0 (0) | 1 (1)
OSTEOMYELITIS (Infections and infestations) | 1 (1) | 1 (1)
OTITIS MEDIA (Infections and infestations) | 4 (4) | 3 (3)
OTITIS MEDIA BACTERIAL (Infections and infestations) | 0 (0) | 1 (1)
PARAINFLUENZAE VIRUS INFECTION (Infections and infestations) | 2 (2) | 0 (0)
PERTUSSIS (Infections and infestations) | 2 (2) | 0 (0)
PHARYNGITIS (Infections and infestations) | 1 (1) | 0 (0)
PHARYNGOTONSILLITIS (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 31 (31) | 27 (28)
PNEUMONIA ADENOVIRAL (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA BACTERIAL (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA BORDETELLA (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA INFLUENZAL (Infections and infestations) | 3 (4) | 0 (0)
PNEUMONIA PARAINFLUENZAE VIRAL (Infections and infestations) | 3 (4) | 1 (1)
PNEUMONIA RESPIRATORY SYNCYTIAL VIRAL (Infections and infestations) | 10 (10) | 2 (2)
PNEUMONIA VIRAL (Infections and infestations) | 1 (1) | 3 (3)
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 0 (0) | 1 (1)
PYELONEPHRITIS (Infections and infestations) | 1 (1) | 2 (2)
PYELONEPHRITIS ACUTE (Infections and infestations) | 0 (0) | 1 (1)
RESPIRATORY SYNCYTIAL VIRUS BRONCHIOLITIS (Infections and infestations) | 40 (43) | 25 (25)
RESPIRATORY SYNCYTIAL VIRUS INFECTION (Infections and infestations) | 3 (3) | 3 (3)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2) | 0 (0)
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 1 (1) | 1 (1)
RHINITIS (Infections and infestations) | 3 (3) | 1 (1)
ROTAVIRUS INFECTION (Infections and infestations) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 2 (2) | 2 (2)
SINUSITIS (Infections and infestations) | 0 (0) | 1 (1)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 (0) | 1 (1)
TRACHEITIS (Infections and infestations) | 2 (3) | 0 (0)
TRACHEOBRONCHITIS (Infections and infestations) | 2 (2) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 22 (23) | 14 (14)
URINARY TRACT INFECTION (Infections and infestations) | 7 (7) | 10 (10)
URINARY TRACT INFECTION BACTERIAL (Infections and infestations) | 2 (2) | 1 (1)
URINARY TRACT INFECTION ENTEROCOCCAL (Infections and infestations) | 1 (1) | 1 (1)
URINARY TRACT INFECTION PSEUDOMONAL (Infections and infestations) | 0 (0) | 1 (1)
UROSEPSIS (Infections and infestations) | 0 (0) | 1 (1)
VARICELLA (Infections and infestations) | 2 (2) | 0 (0)
VIRAL INFECTION (Infections and infestations) | 7 (7) | 4 (4)
VIRAL RHINITIS (Infections and infestations) | 0 (0) | 1 (1)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2) | 6 (7)
WOUND INFECTION (Infections and infestations) | 0 (0) | 1 (2)
CHILD MALTREATMENT SYNDROME (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
DEVICE MALFUNCTION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
FACE INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
FEEDING TUBE COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
FOREIGN BODY TRAUMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HAIR-THREAD TOURNIQUET SYNDROME (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
HEAD INJURY (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
MEDICAL DEVICE COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
POST PROCEDURAL DISCHARGE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
SHUNT MALFUNCTION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SKULL FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
TRAUMATIC BRAIN INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
VENTRICULOPERITONEAL SHUNT MALFUNCTION (Injury, poisoning and procedural complications) | 4 (4) | 2 (3)
VIIITH NERVE INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
BIOPSY RECTUM (Investigations) | 0 (0) | 1 (1)
BLOOD BILIRUBIN INCREASED (Investigations) | 1 (1) | 0 (0)
CYSTOGRAM (Investigations) | 0 (0) | 1 (1)
FALSE POSITIVE LABORATORY RESULT (Investigations) | 0 (0) | 1 (1)
HEPATIC ENZYME INCREASED (Investigations) | 0 (0) | 1 (1)
INVESTIGATION (Investigations) | 1 (1) | 0 (0)
LIVER FUNCTION TEST ABNORMAL (Investigations) | 2 (2) | 0 (0)
MEDICAL OBSERVATION (Investigations) | 1 (1) | 2 (2)
NEUROLOGICAL EXAMINATION (Investigations) | 2 (2) | 1 (1)
OESOPHAGEAL PH (Investigations) | 0 (0) | 1 (1)
OXYGEN SATURATION DECREASED (Investigations) | 2 (5) | 0 (0)
PHYSICAL EXAMINATION (Investigations) | 3 (3) | 3 (3)
WEIGHT DECREASED (Investigations) | 2 (2) | 0 (0)
ANOREXIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
COW'S MILK INTOLERANCE (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 6 (6) | 5 (8)
FEEDING DISORDER OF INFANCY OR EARLY CHILDHOOD (Metabolism and nutrition disorders) | 7 (7) | 2 (3)
FLUID INTAKE REDUCED (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
FLUID OVERLOAD (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERNATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
LACTOSE INTOLERANCE (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
MALNUTRITION (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
WEIGHT GAIN POOR (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
ZINC DEFICIENCY (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
CRANIOSYNOSTOSIS (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
MUSCLE CONTRACTURE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OSTEOPENIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
HAEMANGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 4 (7)
ALTERED STATE OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 1 (1)
CEREBRAL VENTRICLE DILATATION (Nervous system disorders) | 0 (0) | 1 (1)
CONVULSION (Nervous system disorders) | 4 (5) | 3 (5)
CONVULSION NEONATAL (Nervous system disorders) | 1 (2) | 0 (0)
ENCEPHALITIS (Nervous system disorders) | 0 (0) | 1 (1)
EPILEPSY (Nervous system disorders) | 0 (0) | 1 (1)
FEBRILE CONVULSION (Nervous system disorders) | 0 (0) | 1 (1)
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 0 (0) | 1 (2)
HYDROCEPHALUS (Nervous system disorders) | 2 (2) | 5 (5)
HYPERTONIA (Nervous system disorders) | 0 (0) | 1 (1)
HYPOXIC ENCEPHALOPATHY (Nervous system disorders) | 3 (4) | 4 (6)
INTRACRANIAL PRESSURE INCREASED (Nervous system disorders) | 1 (1) | 0 (0)
LETHARGY (Nervous system disorders) | 0 (0) | 2 (3)
MYOCLONUS (Nervous system disorders) | 0 (0) | 1 (1)
SOMNOLENCE (Nervous system disorders) | 1 (1) | 0 (0)
SYNCOPE VASOVAGAL (Nervous system disorders) | 1 (1) | 0 (0)
VOCAL CORD PARESIS (Nervous system disorders) | 0 (0) | 1 (1)
BREATH HOLDING (Psychiatric disorders) | 2 (2) | 0 (0)
RESTLESSNESS (Psychiatric disorders) | 0 (0) | 1 (1)
URETERIC STENOSIS (Renal and urinary disorders) | 1 (1) | 0 (0)
BALANITIS (Reproductive system and breast disorders) | 1 (1) | 0 (0)
OVARIAN CYST (Reproductive system and breast disorders) | 0 (0) | 1 (1)
SCROTAL OEDEMA (Reproductive system and breast disorders) | 1 (1) | 0 (0)
APNOEA (Respiratory, thoracic and mediastinal disorders) | 17 (23) | 14 (16)
APPARENT LIFE THREATENING EVENT (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 7 (7)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
BRONCHIAL HYPERREACTIVITY (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 7 (7)
BRONCHOPNEUMOPATHY (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
BRONCHOPULMONARY DYSPLASIA (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 9 (11)
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (5)
CHOKING (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
FOREIGN BODY ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
HYPOVENTILATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
LARYNGEAL OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
LARYNGEAL STENOSIS (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
LARYNGOSPASM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
LUNG CONSOLIDATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OBSTRUCTIVE AIRWAYS DISORDER (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
PHARYNGEAL INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
PULMONARY CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 2 (2)
PULMONARY HYPERTENSIVE CRISIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
RESPIRATORY DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (4)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
STATUS ASTHMATICUS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
STRIDOR (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
TACHYPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
TONSILLAR HYPERTROPHY (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
VOCAL CORD DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (7)
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
PETECHIAE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
URTICARIA (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
SOCIAL STAY HOSPITALISATION (Social circumstances) | 2 (2) | 4 (4)
VICTIM OF CHILD ABUSE (Social circumstances) | 0 (0) | 1 (1)
CENTRAL VENOUS CATHETERISATION (Surgical and medical procedures) | 0 (0) | 1 (1)
COLOSTOMY CLOSURE (Surgical and medical procedures) | 1 (1) | 0 (0)
EAR TUBE INSERTION (Surgical and medical procedures) | 1 (1) | 0 (0)
GASTROSTOMY CLOSURE (Surgical and medical procedures) | 0 (0) | 1 (1)
GASTROSTOMY TUBE INSERTION (Surgical and medical procedures) | 0 (0) | 1 (1)
ILEOSTOMY CLOSURE (Surgical and medical procedures) | 3 (3) | 0 (0)
NUTRITIONAL SUPPORT (Surgical and medical procedures) | 1 (1) | 0 (0)
VENTRICULO-PERITONEAL SHUNT (Surgical and medical procedures) | 0 (0) | 1 (1)
HAEMORRHAGE (Vascular disorders) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 2 (4) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Palivizumab (N=3298) | Motavizumab (N=3315)
ANAEMIA (Blood and lymphatic system disorders) | 73 (75) | 66 (67)
DACRYOSTENOSIS CONGENITAL (Congenital, familial and genetic disorders) | 33 (34) | 35 (37)
CONJUNCTIVITIS (Eye disorders) | 251 (285) | 246 (271)
ABDOMINAL PAIN (Gastrointestinal disorders) | 70 (73) | 54 (55)
CONSTIPATION (Gastrointestinal disorders) | 227 (262) | 234 (265)
DIARRHOEA (Gastrointestinal disorders) | 274 (306) | 254 (295)
FLATULENCE (Gastrointestinal disorders) | 119 (135) | 126 (170)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 190 (198) | 190 (197)
TEETHING (Gastrointestinal disorders) | 282 (408) | 299 (417)
UMBILICAL HERNIA (Gastrointestinal disorders) | 63 (63) | 77 (77)
VOMITING (Gastrointestinal disorders) | 164 (179) | 158 (174)
INJECTION SITE ERYTHEMA (General disorders) | 28 (38) | 41 (52)
INJECTION SITE PAIN (General disorders) | 49 (94) | 45 (81)
IRRITABILITY (General disorders) | 164 (243) | 193 (299)
PYREXIA (General disorders) | 556 (729) | 543 (718)
BRONCHIOLITIS (Infections and infestations) | 222 (263) | 193 (226)
BRONCHITIS (Infections and infestations) | 260 (356) | 230 (328)
CANDIDIASIS (Infections and infestations) | 79 (93) | 58 (65)
IMMUNISATION REACTION (Immune system disorders) | 97 (122) | 102 (138)
GASTROENTERITIS (Infections and infestations) | 207 (223) | 199 (212)
GASTROENTERITIS VIRAL (Infections and infestations) | 32 (36) | 40 (40)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 133 (165) | 130 (159)
NASOPHARYNGITIS (Infections and infestations) | 262 (333) | 240 (325)
ORAL CANDIDIASIS (Infections and infestations) | 107 (120) | 101 (113)
OTITIS MEDIA (Infections and infestations) | 418 (565) | 432 (575)
OTITIS MEDIA ACUTE (Infections and infestations) | 54 (79) | 65 (83)
PHARYNGITIS (Infections and infestations) | 91 (101) | 70 (81)
PNEUMONIA (Infections and infestations) | 35 (39) | 15 (15)
RHINITIS (Infections and infestations) | 444 (593) | 440 (600)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 981 (1482) | 956 (1420)
VIRAL INFECTION (Infections and infestations) | 98 (112) | 86 (103)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 60 (64) | 56 (64)
BLOOD UREA INCREASED (Investigations) | 25 (25) | 35 (35)
HAEMANGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 38 (41) | 29 (34)
AGITATION (Psychiatric disorders) | 47 (61) | 35 (51)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 37 (45) | 33 (37)
BRONCHIAL HYPERREACTIVITY (Respiratory, thoracic and mediastinal disorders) | 54 (62) | 44 (48)
COUGH (Respiratory, thoracic and mediastinal disorders) | 216 (262) | 220 (260)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 265 (326) | 269 (318)
RESPIRATORY DISORDER (Respiratory, thoracic and mediastinal disorders) | 275 (374) | 295 (380)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 92 (112) | 99 (124)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 70 (85) | 51 (61)
DERMATITIS ATOPIC (Skin and subcutaneous tissue disorders) | 53 (55) | 44 (48)
DERMATITIS DIAPER (Skin and subcutaneous tissue disorders) | 192 (233) | 177 (199)
DRY SKIN (Skin and subcutaneous tissue disorders) | 25 (26) | 35 (37)
ECZEMA (Skin and subcutaneous tissue disorders) | 95 (100) | 132 (140)
RASH (Skin and subcutaneous tissue disorders) | 103 (110) | 130 (147)
SEBORRHOEIC DERMATITIS (Skin and subcutaneous tissue disorders) | 52 (53) | 56 (57)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.